CLINICAL TRIAL: NCT03166475
Title: Ridge Preservation With Provisional Ovoid Pontic: a Randomized and Controlled Clinical-tomographic Trial
Brief Title: Ridge Preservation With Provisional Ovoid Pontic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Bruno Salles Sotto-Maior, Clinical Professor Bruno Salles Sotto-Maior, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reabilitação Oral
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Alveolar Process Atrophy
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Palatal pedicle flap (Group 1) (Experimental): On patients of this group were performed the palatal pedicle subepithelial connective tissue flap after the extraction, following the technique described by Khoury & Happe (2000), which consists of total detachment of the palatal flap followed by division of the flap to release the connective tissue, maintain a pedicle and sliding it to cover the fresh socket by primary intention. The sutures were removed seven to ten days of postoperative.
  Interventions: Procedure: Surgical procedures
- Graft + palatal pedicle flap (Group 2) (Experimental): On patients of this group were performed the palatal pedicle flap like the group 1, however, the sockets were previously filled with a graft of synthetic bone substitute (Bone Ceramic®, Straumann, Switzerland) and then recovered with the connective flap and sutured by primary intention. The sutures were removed seven to ten days of postoperative.
  Interventions: Procedure: Surgical procedures
- Provisional ovoid pontic (Group 3) (Experimental): On patients of this group, after the extraction of the tooth, were made a provisional ovoid pontic with acrylic resin or with the crown of the removed tooth itself, cut and sealed with composite resin. The pontics were placed to seal the entire gingival margin of the socket and penetrating 2 to 3 mm into it, stabilized laterally by the adjacent teeth with orthodontic and composite resin or acrylic resin. No sutures were made.
  Interventions: Procedure: Surgical procedures

INTERVENTIONS:
Procedure: Surgical procedures — All the extractions were performed under local anaesthesia, minimally traumatic as possible. After the extraction, each patient was treated according to the group of their allocations.

SUMMARY:
A prospective randomized controlled trial of 30 patients from the Faculty of Dentistry of the UFJF was conducted. It was included patients who presented indication of extraction of premolars, canines or incisors. All the thirty patients underwent dental extraction and were randomly divided into three groups according to the study methodology. Plaster casts and Cone-Beam Computed Tomography (CBCT) exams were performed for comparative analysis between sample groups and between study times ( imediate postoperative and four months later).

DETAILED DESCRIPTION:
Thirty consecutive patients who presented at the Dentistry College of Federal University of Juiz de Fora (Brazil) were selected, requiring a single-tooth extraction of premolar, canines or incisors in maxilla. All of the patients included at this study signed a free and informed consent form, agreeing to participate voluntarily in this research. The study was approved by the Research Ethical Committee of the University of Juiz de Fora under the form 1.731.395.

The patients were randomly allocated in three groups according the following treatments:

* Group 1: Closure of the socket by primary intention through a palatal pedicle subepithelial connective tissue flap by the technique of Khoury & Happe (2000) (Figure 1);
* Group 2: Filling the socket with a synthetic bone substitute of biphasic calcium phosphate (Bone Ceramic®, Straumann) and covering it with a palatal pedicle flap by the technique of Khoury & Happe (2000) (Figure 2);
* Group 3: Sealing of the socket with a provisional ovoid pontic of acrylic resin (Figure 3).

As response factors were performed evaluations of study casts and tomographic analysis for dimensional stability evaluation of the sockets at immediate postoperative and after four months of the surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of extraction of premolars, canines or incisors, which has two adjacent teeth, due to root fracture, extensive caries that did not allow unfavorable restorative and / or endodontic prognosis, systemically healthy.

Exclusion Criteria:

* Patients who use any drug that influences bone metabolism, patients with a history of head radiotherapy and neck, patients undergoing chemotherapy for the treatment of malignant tumors at the time of the study, patients with socket severely reabsorbed, smokers and pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Changes of bone remodelation measured by Cone-Beam Computed Tomography exams and by plaster casts analysis, from baseline to 4 months | Baseline (immediate postoperative) and 4 months after it.
  Will be measured width and height buccal-lingual of the ridge for each tooth extracted by the researcher.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers, the data will be used for the same researcher on other research later.

REFERENCES:
- [Result] Ten Heggeler JM, Slot DE, Van der Weijden GA. Effect of socket preservation therapies following tooth extraction in non-molar regions in humans: a systematic review. Clin Oral Implants Res. 2011 Aug;22(8):779-88. doi: 10.1111/j.1600-0501.2010.02064.x. Epub 2010 Nov 22. PMID 21091540
- [Result] Iocca O, Farcomeni A, Pardinas Lopez S, Talib HS. Alveolar ridge preservation after tooth extraction: a Bayesian Network meta-analysis of grafting materials efficacy on prevention of bone height and width reduction. J Clin Periodontol. 2017 Jan;44(1):104-114. doi: 10.1111/jcpe.12633. Epub 2016 Dec 5. PMID 27712001
- [Result] Nevins M, Camelo M, De Paoli S, Friedland B, Schenk RK, Parma-Benfenati S, Simion M, Tinti C, Wagenberg B. A study of the fate of the buccal wall of extraction sockets of teeth with prominent roots. Int J Periodontics Restorative Dent. 2006 Feb;26(1):19-29. PMID 16515093
- [Result] Araujo MG, da Silva JCC, de Mendonca AF, Lindhe J. Ridge alterations following grafting of fresh extraction sockets in man. A randomized clinical trial. Clin Oral Implants Res. 2015 Apr;26(4):407-412. doi: 10.1111/clr.12366. Epub 2014 Mar 12. PMID 24621203
- [Result] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Result] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Relationship between the buccal bone plate thickness and the healing of postextraction sockets with/without ridge preservation. Int J Periodontics Restorative Dent. 2014 Mar-Apr;34(2):211-7. doi: 10.11607/prd.1885. PMID 24600657
- [Result] Nart J, Barallat L, Jimenez D, Mestres J, Gomez A, Carrasco MA, Violant D, Ruiz-Magaz V. Radiographic and histological evaluation of deproteinized bovine bone mineral vs. deproteinized bovine bone mineral with 10% collagen in ridge preservation. A randomized controlled clinical trial. Clin Oral Implants Res. 2017 Jul;28(7):840-848. doi: 10.1111/clr.12889. Epub 2016 Jun 22. PMID 27335267
- [Result] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Result] Khoury F, Happe A. The palatal subepithelial connective tissue flap method for soft tissue management to cover maxillary defects: a clinical report. Int J Oral Maxillofac Implants. 2000 May-Jun;15(3):415-8. PMID 10874807
- [Result] Mardas N, Chadha V, Donos N. Alveolar ridge preservation with guided bone regeneration and a synthetic bone substitute or a bovine-derived xenograft: a randomized, controlled clinical trial. Clin Oral Implants Res. 2010 Jul;21(7):688-98. doi: 10.1111/j.1600-0501.2010.01918.x. PMID 20636724
- [Result] Ryu KH, Min S, You HK, Sin YW, Lee W, Lee J, Kiss A, Almohaimeed M, Zadeh HH. Alveolar ridge dimensional changes following ridge preservation procedure using SocketKAP() : exploratory study of serial cone-beam computed tomography and histologic analysis in canine model. Clin Oral Implants Res. 2016 Sep;27(9):1144-51. doi: 10.1111/clr.12711. Epub 2015 Dec 13. PMID 26660705
- [Result] Fickl S, Fischer K, Petersen N, Happe A, Schlee M, Schlagenhauf U, Kebschull M. Dimensional Evaluation of Different Ridge Preservation Techniques: A Randomized Clinical Study. Int J Periodontics Restorative Dent. 2017 May/Jun;37(3):403-410. doi: 10.11607/prd.2629. PMID 28402351